CLINICAL TRIAL: NCT02340676
Title: A Phase II Trial of Low-Dose Interleukin-2 (IL-2) Added to Extra-Corporeal Photopheresis for Steroid-Refractory Chronic Graft-versus-Host-Disease
Brief Title: A Phase II Trial of Low-Dose Interleukin-2 (IL-2) Added to Extra-Corporeal Photopheresis for Steroid-Refractory cGVHD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-479
Record Dates: First submitted 2015-01-07; First posted 2015-01-19 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: chronic graft-versus-host-disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Photopheresis; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ECP plus IL-2 (Experimental): * Extracorporeal Photopheresis (ECP) standard-of-care
  * Daily subcutaneous (SC) interleukin-2 (IL-2) (Proleukin®) during predetermined weeks of treatment cycle
  Interventions: Procedure: Extracorporeal Photopheresis (ECP); Drug: Interleukin-2

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis (ECP) — Participants receive ECP treatment twice a week for 16 weeks
Drug: Interleukin-2 — Participants receive daily IL-2 injections starting Week 8 of study and ending at Week 16
  Other Names: IL-2; Proleukin®

SUMMARY:
This research study is evaluating a combination of a therapy called Extra-corporeal Photopheresis (ECP) with a drug called Interleukin-2 (IL-2) as a possible treatment for chronic graft-versus-host-disease (GVHD) following allogeneic stem cell transplant.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved IL-2 for the treatment of chronic GVHD but it has been approved for metastatic renal cell carcinoma (MCC) and metastatic melanoma. ECP is a standard of care treatment for chronic GVHD that has not responded to steroids.

Chronic GVHD is a medical condition that may occur after receiving bone marrow, stem cell or cord blood transplant from a donor. The donor's immune system may recognize (the host) as foreign and attempt to 'reject' it. This process is known as graft-versus-host disease.

Traditional standard therapy to treat chronic GVHD is prednisone (steroids). Participants on this trial have not responded to steroid therapy. The investigstors are looking to assess whether the combination of IL-2 and ECP therapy helps control chronic GVHD by stopping the donor's immune system from 'rejecting' the participant's body.

Participants will receive standard-of-care ECP treatment two times a week for 16 weeks. Each treatment will last approximately 2-3 hours. Starting after Week 8 of the ECP treatments, participants will give themselves or be given IL-2 through an injection under their skin. Participants will do this once every day for 8 weeks until the end of the 16-week ECP treatment. If a participant's GVHD worsens during the initial 8 weeks of ECP treatment, he or she has the option of starting IL-2 early.

If a participant's chronic GVHD improves at the end of the 16-week study duration, he or she may have the option of continuing the combination therapy of ECP and IL-2. Extended duration therapy is twice weekly ECP treatments plus daily IL-2 starting at the end of week 16. Participants may also have the option of continuing ECP treatments without IL-2 after the end of Week 16. If this is the case, participants will only be followed for one year from the start of therapy and will not have required study visits or tests.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

* Recipients of 7-8/8 HLA matched adult donor allogeneic stem cell transplantation with myeloablative or non-myeloablative conditioning regimens.
* Participants must have steroid-refractory cGVHD. Steroid-refractory cGVHD is defined as having persistent signs and symptoms of cGVHD (Appendix D; section 17.4) despite the use of prednisone at ≥ 0.25 mg/kg/day (or 0.5 mg/kg every other day) for at least 4 weeks (or equivalent dosing of alternate corticosteroids) without complete resolution of signs and symptoms. Patients with either extensive chronic GVHD or limited chronic GVHD requiring systemic therapy are eligible.
* Stable dose of corticosteroids for 4 weeks prior to enrollment
* No addition or subtraction of other immunosuppressive medications (e.g., calcineurin-inhibitors, sirolimus, mycophenolate-mofetil) for 4 weeks prior to enrollment. The dose of immunosuppressive medicines may be adjusted based on the therapeutic range of that drug
* Patient age ≥18 years old. Because no dosing or adverse event data are currently available on the use of IL-2 in participants <18 years of age, children are excluded from this study.
* Estimated life expectancy greater than 3 months.
* ECOG performance status 0-2 (Appendix A; section 17.1).
* Participants must have adequate organ function as defined below:

  * Hepatic: Adequate hepatic function (total bilirubin <2.0 mg/dl-exception permitted in patients with Gilbert's Syndrome; AST (SGOT)/ALT (SGPT) ≤ 2x ULN), unless hepatic dysfunction is a manifestation of presumed cGVHD. For patients with abnormal LFTs as the sole manifestation of cGVHD, documented GVHD on liver biopsy will be required prior to enrollment. Abnormal LFTs in the context of active cGVHD involving other organ systems may also be permitted if the treating physician documents the abnormal LFTs as being consistent with hepatic cGVHD, and a liver biopsy will not be mandated in this situation.
  * Renal: Serum creatinine within normal institutional limits or creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
  * Pulmonary: FEV1 ≥ 50% or DLCO(Hb) ≥ 40% of predicted, unless pulmonary dysfunction is deemed to be due to chronic GVHD.
  * Adequate bone marrow function indicated by ANC>1000/mm3 and platelets>50,000/mm3 without growth factors or transfusions
  * Cardiac: No myocardial infarction within 6 months prior to enrollment or NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* The effects of IL-2 on the developing human fetus are unknown. For this reason and because chemotherapeutic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

* Ongoing prednisone requirement >1 mg/kg/day (or equivalent).
* Concurrent use of calcineurin-inhibitors plus sirolimus. Either agent alone is acceptable.
* History of thrombotic microangiopathy, hemolytic-uremic syndrome or thrombotic thrombocytopenic purpura.
* Exposure to any new immunosuppressive medication in the 4 weeks prior to enrollment.
* Extra-corporeal Photopheresis (ECP) or rituximab therapy within 4 weeks prior to enrollment
* Any contraindication to ECP, i.e. contraindication to heparin or 8-MOP.
* Post-transplant exposure to any novel immunosuppressive medication (e.g., alemtuzumab) within 100 days prior to enrollment.
* Donor lymphocyte infusion within 100 days prior to enrollment.
* Active malignant relapse.
* Active uncontrolled infection.
* Inability to comply with IL-2 treatment regimen.
* Uncontrolled cardiac angina or symptomatic congestive heart failure (NYHA Class III or IV: Appendix C; section 17.3).
* Organ transplant (allograft) recipient.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the agents used after allogeneic HSCT. In addition, these individuals are at increased risk of lethal infections. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Individuals with active hepatitis B or C are ineligible as they are at high risk of lethal treatment-related hepatotoxicity after HSCT.
* Other investigational drugs within 4 weeks prior to enrollment, unless cleared by the Principal Investigator.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02; Primary Completion 2017-08 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, MBBS,D.Phil, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Insitute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Belizaire R, Kim HT, Poryanda SJ, Mirkovic NV, Hipolito E, Savage WJ, Reynolds CG, Fields MJ, Whangbo J, Kubo T, Nikiforow S, Alyea EP, Armand P, Cutler CS, Ho VT, Blazar BR, Antin JH, Ritz J, Soiffer RJ, Koreth J. Efficacy and immunologic effects of extracorporeal photopheresis plus interleukin-2 in chronic graft-versus-host disease. Blood Adv. 2019 Apr 9;3(7):969-979. doi: 10.1182/bloodadvances.2018029124. PMID 30936057

RESULTS

PARTICIPANT FLOW:
Groups:
- ECP Plus IL-2: * Extracorporeal Photopheresis (ECP) standard-of-care
  * Daily subcutaneous (SC) interleukin-2 (IL-2) (Proleukin®) during predetermined weeks of treatment cycle
  Extracorporeal Photopheresis (ECP): Participants receive ECP treatment twice a week for 16 weeks
  Interleukin-2: Participants receive daily IL-2 injections starting Week 8 of study and ending at Week 16
Period: Overall Study
Arm/Group | ECP Plus IL-2
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ECP Plus IL-2
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 62 [34 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Chronic Graft-versus-Host Disease (cGVHD) [Count of Participants; unit: Participants]
  Mild | 1
  Moderate | 19
  Severe | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participant With Response at Week 16
Description: Participants will have their cGVHD evaluated at baseline through Week 16.
Time Frame: Baseline through Week 16 of the study
Population: 22 evaluable for efficacy
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | ECP Plus IL-2
Number analyzed (Participants) | 25
percentage of patients | 59 [40 to 77]

2. Secondary Outcome: Number of Grade 3 or Higher Toxicities Related to ECP Plus Low-dose SC IL-2 Therapy
Description: All Grade 3 or higher toxicities related to ECP plus low-dose SC IL-2 therapy have been reported.
Time Frame: Baseline through Week 16 of the study
Measure: Number; unit: Occurrance of reported grade
Arm/Group | ECP Plus IL-2
Number analyzed (Participants) | 25
Occurrance of reported grade
  Grade 3 | 5
  Grade 4 | 0
  Grade 5 | 0

3. Secondary Outcome: Regulatory T Cell Counts During ECP Plus Low-dose Daily SC IL-2
Description: Assays will be conducted to detect Change in Regulatory T cell counts during ECP plus low-dose daily SC IL-2
Time Frame: Baseline through Week 16 of the study
Measure: Median (Inter-Quartile Range); unit: cells/uL
Arm/Group | ECP Plus IL-2
Number analyzed (Participants) | 25
cells/uL
  Baseline | 11.7 [5.6 to 18.2]
  Week 16 | 50.7 [32.5 to 75.4]

4. Secondary Outcome: Prednisone Use During ECP Plus Low-dose IL-2 From Baseline Through Week 16 of Study
Description: Prednisone use was assessed during ECP plus low-dose IL-2 treatment at baseline through Week 16 of study.
Time Frame: Baseline through Week 16 of the study
Measure: Median (Full Range); unit: median percentage of change
Arm/Group | ECP Plus IL-2
Number analyzed (Participants) | 25
median percentage of change | 25 [-67 to 300]

5. Secondary Outcome: Overall Survival
Description: Overall survival From the start of treatment to 1 Year was assessed
Time Frame: From the start of treatment to 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | ECP Plus IL-2
Number analyzed (Participants) | 25
percentage of probability | 80 [58 to 91]

6. Secondary Outcome: Progression-free Survival
Description: One year overall survival was analyzed
Time Frame: From the start of treatment to 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | ECP Plus IL-2
Number analyzed (Participants) | 25
percentage of probability | 76 [54 to 88]

7. Secondary Outcome: Non-relapse Mortality
Description: Participants one year cumulative incidence of Non-relapse mortality was assessed.
Time Frame: From the start of treatment to 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | ECP Plus IL-2
Number analyzed (Participants) | 25
percentage of probability | 20 [7 to 38]

8. Secondary Outcome: Relapse at 1 Year
Description: Relapse at 1 year was assessed
Time Frame: From the start of treatment to 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | ECP Plus IL-2
Number analyzed (Participants) | 25
percentage of probability | 4 [0.3 to 17]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from initiation of study intervention, throughout the study, and within 30 days of the last study intervention.
Description: Reporting Participating investigators assessed the occurrence of Adverse Events and Serious Adverse Events at all participant evaluation time points during the study.
Arm/Group | ECP Plus IL-2
All-Cause Mortality (participants affected / at risk) | 3/25
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECP Plus IL-2 (N=25)
Bronchiolitis Obliterans Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 Participant passed away to Grad5 Bronchiolitis Obliterans Syndrome. Expected and unrelated to study treatment.
Parainfluenza Type 3 (Infections and infestations) | 1 (1) — 1 Participant passed away due to Grade 5 Parainfluenza Type 3. Expected and unrelated to study treatment.
Cardiac Arrest (Cardiac disorders) | 1 (1) — 1 Participant passed away to Grade 5 Cardiac Arrest. Unexpected and unrelated to study treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECP Plus IL-2 (N=25)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 Participant experienced Grade 2 Cough. Unexpected and possible to study treatment.
Acute Limb Schemia (Vascular disorders) | 1 (1) — 1 Participant experienced Grade 3 Acute Limb Ischemia. Unexpected and possible to study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT02340676/Prot_SAP_000.pdf